CLINICAL TRIAL: NCT03849820
Title: Open vs Robotic Assisted Partial Nephrectomy
Acronym: OpeRa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment the study was terminated
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OpeRa-2018
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Renal Cancer
Keywords: Robotic-assisted Surgery; Open Surgery; Partial Nephrectomy; minimal invasive surgery; RAS; MIS
MeSH Terms: conditions — Kidney Neoplasms | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic-assisted partial nephrectomy (Active Comparator): da Vinci surgical robotic assisted partial nephrectomy
  Interventions: Device: Robotic-assisted partial nephrectomy
- Open partial nephrectomy (Active Comparator): Open partial nephrectomy surgery
  Interventions: Other: Open partial nephrectomy

INTERVENTIONS:
Device: Robotic-assisted partial nephrectomy — Application of the da Vinci surgical robot to assist the partial nephrectomy
  Other Names: da Vinci, RAS, dVPN
  Arms: Robotic-assisted partial nephrectomy
Other: Open partial nephrectomy — Open surgery to conduct the partial nephrectomy
  Other Names: Open surgery
  Arms: Open partial nephrectomy

SUMMARY:
To demonstrate that Robotic-Assisted partial nephrectomy is superior to Open partial nephrectomy in reducing the number of 30 day post-operative complications (Clavien-Dindo Type I-V) for patients with intermediate to high complexity kidney tumors.

DETAILED DESCRIPTION:
Partial nephrectomy is the surgical removal of a kidney tumor while unaffected tissue remains intact so that the kidney function is maintained as far as possible. The more radical procedure would be the complete removal of the kidney, which is not examined in this trial.

Surgery will be randomized either to an open technique involving a large incision or the robotic assisted technique with a few small incisions (keyhole surgery). With robotic assisted surgery the movements of the surgeon are translated into the movement of the instruments.

It is not clear which of the two procedures, open or robotic assisted, has less complications. It is expected that these are different due to the different level of invasiveness and the level of direct access to the organ. This study aims to show that robotic assisted surgery results in less complications than open surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient with a renal tumor that is a candidate for OPEN surgery and robotic assisted surgery (RAS) partial nephrectomy (PN)
* R.E.N.A.L. score ≥ 7
* eGFR ≥ 50 ml/min/1.73 m²
* Anticoagulation is accepted according to the surgeon's practice

Exclusion Criteria:

* Solitary kidney or functionally solitary kidney
* Prior surgery at the affected kidney excluding endoscopic kidney stone surgery
* Bilateral tumors
* Multiple renal tumors requiring excision
* Renal vein tumor thrombus
* Likely insufficient volume of remaining parenchyma after partial nephrectomy to maintain viable kidney remnant
* Metastatic disease with life expectancy of less than 1 year
* Pregnancy or suspected pregnancy
* Planned concomitant procedure
* Subject who is unable or unwilling to comply with the protocol requirements
* Subject considered to be from a vulnerable population according to IS0 14155:2011

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
30 day complications | Day of surgery to 30th post operative day
  Any complication that occurred within 30 days post surgery

SECONDARY OUTCOMES:
Operative time | Day of surgery
  Timing of surgical steps in the OR
Ischemia time | Day of surgery
  Period in which the kidney has no blood supply
Surgical radicality conversions | Day of surgery
  Conversion from robotic to open, partial to radical
Intraoperative blood loss | Day of surgery
  Volume of blood loss during the surgical procedure
Pain assessment | Baseline until Day 90
  Assessment of pain level via the Brief Pain Inventory (BPI)
Pain Medication | Baseline until Day 90
  Recording pain medication
Neuropathic pain | Baseline and Day 30 and Day 90
  Development of neuropathic pain via the DN-4 Patient interview questions
Kidney function via the estimated glomerular filtration rate (eGRF) | Baseline until Day 5 / discharge (whatever is earlier)
  Data will be gathered from routine examination, not a mandatory assessment
Post operative complications | Day 90
  Any Clavien-Dindo I-V post-operative complication
Length of stay | Discharge
  Time from surgery to discharge
Procedure related readmissions | Day 90
  Readmission that can be linked to the partial nephrectomy
Procedure related reoperations | Day 90
  Re-operation that can be linked to the partial nephrectomy
Quality of recovery from the intervention | Baseline until Day 5 / discharge (whatever is earlier)
  Quality of recovery questionnaire QoR-9
Quality of life questionnaire, generic measure | Baseline until Day 90
  EQ-5D 5L
Quality of life questionnaire, cancer patient specific | Baseline until Day 90
  EORTC QLQ-C30
Overall survival | Day of surgery to 5 years
  time from surgery to death from any cause
Disease specific survival | Day of surgery to 5 years
  time from surgery to death due to kidney cancer
Disease free survival | Day of surgery to 5 years
  time from surgery to first documented recurrence of renal cell carcinoma as defined by the investigator
Local recurrence free survival | Day of surgery to 5 years
  Time from surgery to the first documented local recurrence e.g. tumor in the operated kidney or in the immediate vicinity (e.g. perirenal fat) at the surgical site. Portside recurrence / incisional, surgical access site recurrence to the affected kidney would also be considered as a local recurrence.
Comprehensive Complication Index | Day of surgery to 30th post operative day
  Any complication that occurred within 30 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc O Grimm, MD, Prof, Principal Investigator — Department of Urology, University Hospital Jena; Arnulf Stenzl, MD, Prof, Principal Investigator — Dept. of Urology, University Hospital Tübingen, Germany
Locations (12):
- Germany (12):
  - Dept. of Urology, University Hospital Tübingen, Tübingen, Germany
  - Department of Urology, University Hospital Düsseldorf, Düsseldorf
  - Department of Urology, Alfried Krupp Krankenhaus Rüttenscheid, Essen
  - Department of Urology, University Hospital Freiburg, Freiburg im Breisgau
  - Universitätsklinik und Poliklinik für Urologie, Halle
  - Universitätsklinikum Heidelberg, Urologische Klinik, Heidelberg
  - Klinik für Urologie, Marien Hospital Herne, Herne
  - Department of Urology - Universitätsklinikum des Saarlandes, Homburg
  - Department of Urology, University Hospital Jena, Jena
  - Klinik für Urologie, Marien-Hospital Marl, Marl
  - Department of Urology, Klinikum rechts der Isar der Technischen Universität, Munich
  - Helios Universitätsklinkum Wuppertal - Department of Urology, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimm MO, Bedke J, Nyarangi-Dix J, Khoder W, Foller S, Sommerfeld HJ, Giessing M, Heck M, Meissner W, Slee A, Leucht K, von Rundstedt F, Theil G, Buse S, Siemer S, Albers P, Gratzke C, Hohenfellner M, Stenzl A. Open versus robotic-assisted partial nephrectomy in patients with intermediate/high-complexity kidney tumours: final results of the randomised, controlled, open-label, multicentre trial OpeRa. Ann Oncol. 2025 Aug;36(8):988-998. doi: 10.1016/j.annonc.2025.04.005. Epub 2025 Apr 16. PMID 40250528